CLINICAL TRIAL: NCT04614103
Title: A Phase 2 Multicenter Study of Autologous Tumor Infiltrating Lymphocytes (TIL or LN-145) in Patients With Metastatic Non-Small-Cell Lung Cancer
Brief Title: Autologous LN-145 in Patients With Metastatic Non-Small-Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Iovance Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-LUN-202; 2020-003629-45 (EudraCT Number); 2024-510778-26-00 (EU CTIS Number)
Record Dates: First submitted 2020-10-21; First posted 2020-11-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: LN-145; Cell Therapy; Autologous Adoptive Cell Therapy; Cellular Immuno-therapy; Tumor Infiltrating Lymphocytes; TIL; IL-2; Non Small Cell Lung Cancer; NSCLC; Second line Lung Cancer; Bronchial Neoplasms; Carcinoma; Lung Disease; Metastatic Lung Cancer; Metastatic Non Small Cell Lung Cancer; Metastatic NSCLC; Lung Carcinoma; PD-L1; Stage IV Lung Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IV NSCLC; Systemic Therapy; 2nd line therapy; Second line therapy; CPI; Immune checkpoint inhibitor (ICI); NSCLC Recurrent; Recurrent Lung Cancer; Recurrent Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms; Carcinoma; Lung Diseases; Lung Neoplasms | interventions — Toll-Like Receptor 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Patients whose tumors did not express programmed cell death-ligand 1 (PD-L1), i.e., tumor proportion score (TPS) < 1% prior to ICI treatment and Patients with no available historical TPS for PD-L1 expression
  Interventions: Biological: LN-145
- Cohort 2 (Experimental): Patients whose tumors expressed PD-L1 TPS ≥1% prior to ICI treatment
  Interventions: Biological: LN-145
- Cohort 3 (Experimental): Patients, regardless of tumor PD-L1 TPS prior to ICI treatment, who are unable to safely undergo a surgical tumor resection for TIL generation
  Interventions: Biological: LN-145
- Cohort 4 (Experimental): Patients, regardless of tumor PD-L1 expression status prior to ICI treatment, who have meet all inclusion/exclusion criteria except the requirement to have documented disease progression may elect to have the tumor harvest procedure and TIL production prior to disease progression on their current anticancer treatment. Documentation of progressive disease and identification of a target lesion for RECIST v1.1 assessment is required at Baseline for these patients.
  Interventions: Biological: LN-145
- Retreatment Cohort (Experimental): Patients who were previously treated with LN-145 in Cohort 1, 2, 3, or 4.
  Interventions: Biological: LN-145

INTERVENTIONS:
Biological: LN-145 — A tumor sample is resected from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepleting chemotherapy including cyclophosphamide and fludarabine, patient is infused with autologous TIL (LN-145), followed by IL-2.
  Other Names: TIL, Autologous Tumor Infiltrating Lymphocytes
  Arms: Cohort 1; Cohort 2; Cohort 4; Retreatment Cohort
Biological: LN-145 — A tumor sample is obtained by image-guided core biopsy from each patient and cultured ex vivo to expand the population of tumor infiltrating lymphocytes. After lymphodepleting chemotherapy including cyclophosphamide and fludarabine, patient is infused with autologous TIL (LN-145) followed by IL-2.
  Other Names: TIL, Autologous Tumor Infiltrating Lymphocytes
  Arms: Cohort 3

SUMMARY:
This is a prospective, open-label, multi-cohort, non-randomized, multicenter phase 2 study evaluating LN-145 in patients with metastatic non-small-cell lung cancer

DETAILED DESCRIPTION:
LN-145 is a ready-to-infuse TIL therapy that utilizes an autologous TIL manufacturing process, as originally developed by the NCI and further optimized by Iovance for the treatment of patients with metastatic NSCLC. The cell transfer therapy used in this study involves patients receiving a non-myeloablative (NMA) lymphodepleting preparative regimen, followed by infusion of autologous TIL, then finally followed by the administration of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 70 years of age may be allowed to enroll after discussion with the Medical Monitor.
* Have historically or pathologically confirmed diagnosis of metastatic Stage IV NSCLC without EGFR, ALK, or ROS1 genomic alterations.
* For patients who have actionable mutations (other than EGFR, ALK, or ROS1 genomic alterations), 1 additional line of therapy with the appropriate health authority approved targeted therapy is required.
* Patients must have documented radiographic disease progression on or after the first-line therapy, including concurrent or sequential ICI and platinum-based chemotherapy ± bevacizumab. No more than 1 prior line is allowed if ICI and platinum-based chemotherapy were administered concurrently and no more than 2 prior lines are allowed for sequential administration of platinum-based chemotherapy and ICI as 2 separate lines.
* LN-145 manufacture is allowed for patients who have residual resectable disease after completion of the platinum-based chemotherapy component of the front-line ICI and platinum-based chemotherapy combination and meet all eligibility criteria except documented disease progression. These patients must intend to receive TIL therapy after disease progression
* Prior systemic therapy in the adjuvant or neoadjuvant setting, or as part of definitive chemoradiotherapy, will count as a line of therapy if the patient had disease progression during or within 12 months after the completion of such therapy.
* At least 1 resectable lesion for TIL production and at least one remaining measurable lesion, as defined by RECIST v1.1
* Have adequate organ function
* LVEF > 45%, NYHA Class 1
* Have adequate pulmonary function
* ECOG performance status of 0 or 1
* Patients of childbearing potential or those with partners of childbearing potential must be willing to practice an approved method of highly effective birth control during treatment and up to 12 months after all protocol-related therapy

Exclusion Criteria:

* Patients who have EGFR, ALK or ROS1 driver mutations
* Patients who have symptomatic, untreated brain metastases.
* Patients who have had allogeneic organ transplant or prior cell therapy within the past 20 years
* Patients who have any form of primary immunodeficiency
* Patients who are on systemic steroid therapy ≥ 10 mg/day of prednisone or equivalent.
* Patients who have received a live or attenuated vaccination within 28 days prior to the start of treatment
* Patients who have had another primary malignancy within the previous 3 years
* Participation in another interventional clinical study within 21 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 60 months
  To evaluate the efficacy of LN-145 as determined by objective response rate (ORR) in patients with metastatic NSCLC using the Response Evaluation Criteria in Solid Tumors (RECIST v1.1), as assessed by central review for Cohorts 1 and 2 and by the investigator for Cohorts 3, 4 and the Retreatment Cohort

SECONDARY OUTCOMES:
Objective Response Rate | Up to 60 months
  To evaluate the efficacy of LN-145 as determined by objective response rate (ORR) per RECIST v1.1, as assessed by the Investigator for Cohorts 1 and 2
Complete Response Rate | Up to 60 months
  To evaluate efficacy parameters such as Complete Response Rate (CRR) per RECIST v1.1
Duration of Response | Up to 60 months
  To evaluate efficacy parameters such as Duration of Response (DOR) rate per RECIST v1.1
Disease Control Rate | Up to 60 months
  To evaluate efficacy parameters such as Disease Control Rate (DCR) per RECIST v1.1
Progression-Free Survival | Up to 60 months
  To evaluate efficacy parameters such as Progression-Free Survival (PFS) per RECIST v1.1
Overall Survival | Up to 60 months
  To evaluate efficacy parameters such as Overall Survival (OS)
Adverse Events | Up to 60 months
  To characterize the safety profile of LN-145 in patients with non-small-cell lung cancer (NSCLC)
Core Biopsies | Up to 60 months
  To determine the feasibility of generating LN-145 using tumor tissue obtained via image-guided core biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Iovance Biotherapeutics Study Team, Study Director — Iovance Biotherapeutics
Locations (84):
- United States (45):
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Christiana Care Health System, Newark, Delaware
  - University of Florida Health Cancer Center, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - University of Kentucky-Markey Cancer Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cooper, Camden, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Novant Health - Charlotte, Charlotte, North Carolina
  - Novant Health - Winston-Salem, Winston-Salem, North Carolina
  - Atrium Health Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Allegheny General Hospital, Natrona Heights, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - Avera Medical Group Cancer Institute, Sioux Falls, South Dakota
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - VCU Medical Center (Virginia Commonwealth University), Richmond, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Hollywood Private Hospital Ramsay, Nedlands, Western Australia
- Canada (2):
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal
  - Princess Margaret Cancer Centre, Toronto
- France (3):
  - Institut Paoli Calmettes, Marseille
  - CHU Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (3):
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Carl Gustav Carus, MK I, Dresden
  - Universitätsklinikum Mannheim, Mannheim
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - IRCCS Fondazione del Piemonte per l'Oncologia, Piemonte
- Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Gachon Unversity Gil Medical Center, Incheon
  - Severance Hospital, Yonsei University, Seoul
- Spain (13):
  - Hospital Universitario A Coruña, A Coruña
  - Instituto Oncologico Rosell, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Clinical Universitaria de Navarra, Pamplona
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois Lausanne, Lausanne, Canton of Vaud
  - University Hospital of Zurich/ Universitätsspital Zürich, Zurich
- United Kingdom (5):
  - Royal Marsden Hospital, Chelsea, England
  - Sarah Cannon Research Institute, London, England
  - University College London, London, England
  - The Christie NHS Foundation Trust, Manchester, England
  - Guy's Hospital, London